CLINICAL TRIAL: NCT02139826
Title: A Randomised, Single-dose, 3-way Crossover Study to Evaluate the Relative Bioavailability of the IX-01 Capsule Formulation Compared With the IX-01 Aqueous Dispersion Formulation, and the Effect of Food on the IX-01 Capsule Formulation, in Healthy Male Subjects
Brief Title: Relative Bioavailability and Food Effect Study of IX-01 Capsules in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ixchelsis Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IX-0102
Record Dates: First submitted 2014-05-12; First posted 2014-05-15 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IX-01 Capsule while Fasting (Experimental): Singe oral dose of 800 milligrams of IX-01 as a capsule, while fasting, in 1 of 3 treatment periods
  Interventions: Drug: IX-01
- IX-01 Aqueous Dispersion while Fasting (Experimental): Single oral dose of 800 milligrams IX-01 as an aqueous dispersion, while fasting in 1 of 3 treatment periods
  Interventions: Drug: IX-01
- IX-01 Capsule after Food (Experimental): Single oral dose of 800 milligrams IX-01 as a capsule, after food, in 1 of 3 treatment periods
  Interventions: Drug: IX-01

INTERVENTIONS:
Drug: IX-01

SUMMARY:
The purpose of this study is to compare the absorption and blood levels of IX-01 when given as a capsule compared to liquid form, and how food affects the absorption in healthy men.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (Quetelet index) in the range 18-30 kilograms/meters squared (kg/m2)
* Body Mass Index = weight [kg] divided by (height [m])2
* Total body weight greater than (>)50 kg at screening
* Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial
* Participants and their partners must be willing to use adequate forms of contraception and to comply with the contraception requirements during the trial and for 4 months after the last dose of medication
* Willingness to give written consent to have data entered into The Over Volunteering Prevention System

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment, including:

  * Lipid and/or liver function test results >1.25 x Upper Limit of Normal (ULN) or other clinical laboratory blood biochemistry test results outside the normal reference range unless discussed and approved by sponsor
  * International normalised ratio (INR) of >1.2 or a platelet count < 150 x 109/Liter
  * History of unexplained syncope
  * Family history of unexplained sudden death, or sudden death due to long QT syndrome
  * Fridericia Correction Formula (QTcF) interval >450 milliseconds (msec) at screening
  * Bundle branch block and other conduction abnormalities, other than mild first degree atrio-ventricular block
  * Irregular rhythms other than sinus arrhythmia or occasional supraventricular ectopic beats
  * T-wave configuration of insufficient quality for determination of QT interval, as assessed by the investigator
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate participation in the trial
* Impaired gastrointestinal, endocrine, thyroid, hepatic, cardiovascular, respiratory, haematological, renal or neurological function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness
* Surgery (for example (e.g.) stomach bypass) or medical condition that might affect absorption, metabolism or elimination of medicines
* Any skin condition, abnormality of the lumbar spine, medical or surgical condition that would preclude lumbar puncture (e.g. coagulopathy, local or systemic infection, left ventricular outflow obstruction, aortic stenosis, previous back surgery)
* Presence or history of severe adverse reaction to any drug
* Use of any prescription or over-the-counter medicine during the 14 days before the first dose of trial medication, or intention to use any medicine during the trial, with the exception of short courses of medication considered by the investigator not to interfere with the safety of the participant or the integrity of the trial data (such as acetaminophen (paracetamol))
* Current use of any herbal remedy or nutritional supplement, or intention to use any such product during the study
* Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months.
* Previous participation in this trial or any other clinical trial of an oxytocin receptor antagonist
* Presence or history of drug or alcohol abuse, or intake of more than 21 units of alcohol weekly or more than 5 cigarettes daily
* Blood pressure and heart rate in supine position at the screening examination outside the ranges 100-130 millimeters of mercury (mm Hg) systolic, 60-90 mm Hg diastolic; heart rate 50-100 beats/minute. Measurements must be made in duplicate, and all values must fall within the acceptable ranges
* Possibility that the participant will not cooperate with the requirements of the protocol
* Evidence of drug abuse on urine testing
* Positive test for hepatitis B, hepatitis C, Human Immunodeficiency Virus 1 (HIV1) or Human Immunodeficiency Virus 2 (HIV2)
* Loss of more than 400 mL blood during the 3 months before the trial, e.g. as a blood donor
* Objection by General Practitioner (GP), on medical grounds, to participant entering trial
* Employee of the investigator site or any company involved in sponsoring, organizing or conducting the trial, or immediate family of the employee

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email: Ixchelsis@Choruspharma.com, Study Director — Ixchelsis Limited
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant withdrew between arms following a non-serious adverse event - unlikely to be treatment-related
Groups:
- Overall Study: Single oral dose of 800 milligrams IX-01 as an aqueous dispersion while fasting, or as a capsule while fasting, or as capsule while fed, in each of 3 treatment periods
  IX-01
Period: Overall Study
Arm/Group | Overall Study
Started | 12
Completed | 11
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All 12 randomized participants
Arm/Group | Overall Study
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12

OUTCOME MEASURES:

1. Primary Outcome: Relative Bioavailability (Frel) of a Capsule Compared to a Liquid Formulation of IX-01 While Fasting, as Calculated by a Ratio of Area Under the Plasma Concentration Time Curve From Time 0 to Infinity
Time Frame: Pre-dose up to 96 hours post dose
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio: capsule fasted/acqueous fasted
Groups:
- IX-01 Capsule While Fasting: Singe oral dose of 800 milligrams of IX-01 as a capsule, while fasting, in 1 of 3 treatment periods
  IX-01
Arm/Group | IX-01 Capsule While Fasting
Number analyzed (Participants) | 11
Ratio: capsule fasted/acqueous fasted | 99.93 [90.8 to 109.98]

2. Primary Outcome: Relative Bioavailability (Frel) of a Capsule Formulation of IX-01 in the Fed State Compared to the Fasted State, as Calculated by a Ratio of Area Under the Plasma Concentration Time Curve From Time 0 to Infinity
Time Frame: Pre-dose up to 96 hours post dose
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio: capsule fed/fasted
Groups:
- IX-01 Capsule After Food: Single oral dose of 800 milligrams IX-01 as a capsule, after food, in 1 of 3 treatment periods
  IX-01
Arm/Group | IX-01 Capsule After Food
Number analyzed (Participants) | 11
Ratio: capsule fed/fasted | 148.85 [135.25 to 163.82]

3. Primary Outcome: Relative Bioavailability (Frel) of a Capsule Compared With a Liquid Formulation of IX-01 While Fasting, as Calculated by a Ratio of Peak Plasma Concentrations
Time Frame: Pre-dose up to 96 hours post dose
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio: capsule/aqueous
Arm/Group | IX-01 Capsule While Fasting
Number analyzed (Participants) | 11
Ratio: capsule/aqueous | 123.78 [96.76 to 158.36]

4. Primary Outcome: Relative Bioavailability (Frel) of a Capsule Formulation of IX-01 in a Fed State Compared to a Fasted State, as Calculated by a Ratio of Peak Plasma Concentrations
Time Frame: Pre-dose up to 96 hours post dose
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio: capsule fed/fasting
Arm/Group | IX-01 Capsule After Food
Number analyzed (Participants) | 11
Ratio: capsule fed/fasting | 175.46 [137.15 to 224.47]

5. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to Infinity, Following a Single Dose of IX-01
Time Frame: Pre-dose and up to 96 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- IX-01 Aqueous Dispersion While Fasting: Single oral dose of 800 milligrams IX-01 as an aqueous dispersion, while fasting in 1 of 3 treatment periods
  IX-01
Arm/Group | IX-01 Aqueous Dispersion While Fasting | IX-01 Capsule While Fasting | IX-01 Capsule After Food
Number analyzed (Participants) | 11 | 11 | 12
h*ng/mL | 20465 (38.9) | 20522 (31.7) | 31613 (27.3)

6. Primary Outcome: Peak Plasma Concentration (Cmax) of IX-01
Time Frame: Pre-dose and up to 96 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | IX-01 Aqueous Dispersion While Fasting | IX-01 Capsule While Fasting | IX-01 Capsule After Food
Number analyzed (Participants) | 11 | 11 | 12
ng/mL | 1147 (39.9) | 1428 (47.9) | 2518.5 (22.7)

7. Primary Outcome: Time to Peak Plasma Concentration (Tmax) of IX-01
Time Frame: Pre-dose up to 96 hours post dose
Measure: Median (Full Range); unit: hours
Arm/Group | IX-01 Aqueous Dispersion While Fasting | IX-01 Capsule While Fasting | IX-01 Capsule After Food
Number analyzed (Participants) | 11 | 11 | 12
hours | 1 [0.5 to 8] | 1.5 [0.75 to 4] | 4 [2 to 8]

8. Primary Outcome: Elimination Half Life (t1/2) of IX-01
Time Frame: Pre-dose up to 96 hours post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | IX-01 Aqueous Dispersion While Fasting | IX-01 Capsule While Fasting | IX-01 Capsule After Food
Number analyzed (Participants) | 11 | 11 | 12
hours | 15 (60.7) | 12.6 (32) | 12.2 (40.2)

9. Primary Outcome: Elimination Rate Constant (Kel) of IX-01
Time Frame: Pre-dose up to 96 hours post last dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | IX-01 Aqueous Dispersion While Fasting | IX-01 Capsule While Fasting | IX-01 Capsule After Food
Number analyzed (Participants) | 11 | 11 | 12
1/h | 0.046 (60.7) | 0.055 (32) | 0.057 (40.2)

10. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to the Time of the Last Measurable Sample of IX-01
Time Frame: Pre-dose to the time of the last measurable sample
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | IX-01 Aqueous Dispersion While Fasting | IX-01 Capsule While Fasting | IX-01 Capsule After Food
Number analyzed (Participants) | 11 | 11 | 12
h*ng/mL | 19529 (34.5) | 20218 (31.1) | 31270 (26.7)

11. Primary Outcome: Concentration of IX-01 in Cerebrospinal Fluid (CSF) After a Single Dose of the Liquid Formulation of IX-01
Description: Listed by time point of 1, 2, 4, 6 hours post dose
Time Frame: 1, 2, 4 and 6 hours after dosing
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IX-01 Aqueous Dispersion While Fasting
Number analyzed (Participants) | 10
ng/mL
  At 1 hour, 1 participant analyzed | 27.8 (0)
  At 2 hours, 2 participants analyzed | 24.4 (2.97)
  At 4 hours, 3 participants analyzed | 54 (17.67)
  At 6 hours, 4 participants analyzed | 40 (21.04)

12. Secondary Outcome: Number of Participants With One or More Drug-Related Adverse Events (AEs) or Any Serious AEs
Time Frame: Baseline to study completion (approximately 6 weeks)
Measure: Number; unit: participants
Arm/Group | IX-01 Aqueous Dispersion While Fasting | IX-01 Capsule While Fasting | IX-01 Capsule After Food
Number analyzed (Participants) | 11 | 11 | 12
participants | 1 | 1 | 2

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Description: The onset date/time of one non-serious event (toothache) was not recorded, so the treatment arm was unknown and not shown below, otherwise all events that occurred during the study period are shown including those that were unrelated
Arm/Group | IX-01 Aqueous Dispersion While Fasting | IX-01 Capsule While Fasting | IX-01 Capsule After Food
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 8/11 | 3/11 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IX-01 Aqueous Dispersion While Fasting (N=11) | IX-01 Capsule While Fasting (N=11) | IX-01 Capsule After Food (N=12)
Procedural Headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (3) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor may choose to collaborate on authorship, and sponsor's agent has 60-day review